CLINICAL TRIAL: NCT01367509
Title: A Phase 1, Open-Label Study to Evaluate Single Dose Pharmacokinetics, Safety, and Tolerability of Methylnaltrexone (MNTX) in Subjects With Impaired Renal Function
Brief Title: Pharmacokinetics, Safety, and Tolerability of Methylnaltrexone (MNTX) in Subjects With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 1105
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): SC Methylnaltrexone (MNTX)
  Interventions: Drug: Methylnaltrexone (MNTX)

INTERVENTIONS:
Drug: Methylnaltrexone (MNTX)

SUMMARY:
This study is evaluating the Pharmacokinetics of MNTX in healthy control subjects and in patients with mild, moderate, or severe renal impairment who do not require hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight >100 lbs. (> 45 kg), and body mass index (BMI) between 18-38 kg/m2, inclusive (BMI 18-30 for the matched reference group)
2. For patients/subjects requiring pharmacotherapy, a stable drug regimen, defined as not having started a new drug or changed dosage within three (3) days or five (5) half-lives (whichever was longer) prior to administration of MNTX concomitant medication must either have conformed to the list of approved drugs and dosage or have been approved by the sponsor.
3. Patients with normal renal function, demographically comparable to the patients with impaired renal function weights and ages were within the range of chronic kidney disease (CKD) group and the average for the matched reference group was within 10 years and 10 kg of the average for the CKD
4. Patients with impaired renal function, good general health except for those illnesses associated with CKD.

Exclusion Criteria:

1. Subjects/patients with any conditions possibly affecting drug absorption (eg. Gastrectomy or clinically significant diabetic gastroenteropathy)
2. Methadone use
3. Consumption of grapefruit or grapefruit juice within seven (7) days prior to administration of study medication.
4. Patients requiring hemodialysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-03; Primary Completion 2005-01 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of MNTX in patients with impaired renal function compared to healthy subjects | 6 days
  To compare the PK of MNTX administered subcutaneously as a single dose in patients with impaired renal function with the PK of MNTX administered to healthy subjects.

SECONDARY OUTCOMES:
Peak time of maximum concentration (Tmax) of MNTX in patients with impaired renal function compared to healthy subjects | 6 days
  To compare the PK of MNTX administered subcutaneously as a single dose in patients with impaired renal function with the PK of MNTX administered to healthy subjects.
Area under the plasma concentration (AUC) of MNTX in patients with impaired renal function compared to healthy subjects | 6 days
  To compare the PK of MNTX administered subcutaneously as a single dose in patients with impaired renal function with the PK of MNTX administered to healthy subjects.
Percent of dose excreted in urine of MNTX in patients with impaired renal function compared to healthy subjects | 6 days
  To compare the PK of MNTX administered subcutaneously as a single dose in patients with impaired renal function with the PK of MNTX administered to healthy subjects.
Urinary clearance of MNTX in patients with impaired renal function compared to healthy subjects | 6 days
  To compare the PK of MNTX administered subcutaneously as a single dose in patients with impaired renal function with the PK of MNTX administered to healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States